CLINICAL TRIAL: NCT02131155
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Afatinib (BIBW 2992) as Adjuvant Therapy After Chemo-radiotherapy in Primary Unresected Patients With Stage III, IVa, or IVb Loco-regionally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: LUX-Head & Neck 4: Afatinib (BIBW 2992) Versus Placebo for the Treatment of Head and Neck Squamous Cell Cancer After Treatment With Chemo-radiotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1200.162
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Afatinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Afatinib (BIBW2992) (Experimental): Once daily
  Interventions: Drug: Afatinib
- Placebo (Placebo Comparator): Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Once daily
  Arms: Placebo
Drug: Afatinib — Once daily
  Arms: Afatinib (BIBW2992)

SUMMARY:
This randomised, double-blind phase III trial will be performed in patients with head and neck squamous cell carcinoma (HNSCC). The objectives of the trial are to compare the efficacy and safety of afatinib (BIBW 2992) with placebo as adjuvant therapy to patients who have received definitive chemo-radiotherapy.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed loco-regionally advanced head and neck squamous cell carcinoma (HNSCC), stage III to IVb
* Unresected tumour prior to chemo-radiotherapy (CRT)
* Concomitant CRT completed prior to randomisation
* After concomitant platinum-based CRT, no evidence of disease (NED) on clinical and radiographic examinations
* Eastern cooperative oncology group (ECOG) performance status 0 or 1

Exclusion criteria:

* Patients with smoking history of less than or equal to 10 pack years and with primary tumour site of base of tongue and/or tonsil
* Cancer of nasopharynx, sinuses, and/or salivary glands
* Prior treatment with epidermal growth factor receptor (EGFR)-targeted small molecules, EGFR-targeted antibodies, and/or any investigational agents for HNSCC
* Known pre-existing Interstitial Lung Disease (ILD)
* Any past or present history of areca/betel-nut chewing or its derivatives for a cumulative duration of more than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (17):
- China (13):
  - 1200.162.86010 Boehringer Ingelheim Investigational Site, Beijing
  - 1200.162.86012 Boehringer Ingelheim Investigational Site, Beijing
  - 1200.162.86019 Boehringer Ingelheim Investigational Site, Changchun
  - 1200.162.86007 Boehringer Ingelheim Investigational Site, Chengdu
  - 1200.162.86017 Boehringer Ingelheim Investigational Site, Fuzhou
  - 1200.162.86005 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1200.162.86003 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1200.162.86013 Boehringer Ingelheim Investigational Site, Jinan
  - 1200.162.86014 Boehringer Ingelheim Investigational Site, Nanning
  - 1200.162.86001 Boehringer Ingelheim Investigational Site, Shanghai
  - 1200.162.86020 Boehringer Ingelheim Investigational Site, Tianjin
  - 1200.162.86004 Boehringer Ingelheim Investigational Site, Wuhan
  - 1200.162.86018 Boehringer Ingelheim Investigational Site, Wuhan
- Singapore, Singapore
- South Korea (2):
  - 1200.162.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.162.82002 Boehringer Ingelheim Investigational Site, Seoul
- 1200.162.88603 Boehringer Ingelheim Investigational Site, Keelung, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib (BIBW2992): Afatinib (BIBW2992) is a film coated tablet. Patients were administered single daily dose of afatinib, starting at 40 milligram (mg) orally with water (~250 millilitre) up to a period of 80 weeks. The dose had to be escalated to 50 mg and/or reduced to 40 mg, 30 mg, or 20 mg.
- Placebo: Single daily dose of matching placebo available for the 50 mg, 40 mg, 30 mg and 20 mg afatinib tablets were administered orally with water (~250 millilitre) up to a period of 80 weeks.
Period: Overall Study
Arm/Group | Afatinib (BIBW2992) | Placebo
Started | 25 (Started are treated patients.) | 11 (Started are treated patients.)
Completed | 0 (Completed are patients who completed study procedures as protocol requires.) | 0 (Completed are patients who completed study procedures as protocol requires.)
Not Completed | 25 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Treatment completed | 1 | 0
Not completed — Primary tumour recurrence | 2 | 1
Not completed — Refused to continue study medication | 1 | 0
Not completed — Study early termination | 20 | 10

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): This analysis set included all patients who were randomised, regardless of taking investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib (BIBW2992) | Placebo | Total
Number analyzed (Participants) | 25 | 11 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (9.70) | 58.4 (6.27) | 56.3 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 25 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS, defined as the number of days from the date of randomisation to the date of tumour recurrence/ Second Primary Tumours (SPT) or death from any cause, whichever occurred first.
  For patients with known date of tumour recurrence/SPT (or death), the event date was the date of tumour recurrence/SPT or the date of death, whichever came first, i.e.
  DFS [day] = minimum (date of tumour recurrence/SPT, date of death) - date of randomisation +1.
  For patients known to be alive and without tumour recurrence/SPT by the end of trial or follow-up visit, they were censored at the date of last imaging when the patient was known to be disease-free and alive:
  DFS (censored) [days] = date of last imaging when the patient was known to be diseasefree and alive - date of randomisation + 1. The Kaplan-Meier (KM) method was to be used to estimate the median DFS for each treatment group. 95% confidence interval (CI) was to be constructed using the Greenwood variance estimate.
Time Frame: up to 4 years
Population: Randomised Set; This study was early terminated and data was available for less than 2/3rds of participants hence per internal Boehringer Ingelheim rules the analysis was not performed as planned in protocol.
Arm/Group | Afatinib (BIBW2992) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Disease Free Survival (DFS) Rate at 2 Years
Description: Disease Free Survival (DFS) rate at 2 years is presented
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Afatinib (BIBW2992) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from the date of randomisation until death.
  For patients with known date of death (regardless of the cause of death):
  OS [days] = date of death - date of randomisation +1
  For patients known to be alive by the end of trial:
  OS (censored) [days] = the last date when the patient was known to be alive - date of randomisation +1 OS was to be analysed similarly to DFS.
Time Frame: up to 4 years
Population: as for outcome 1
Arm/Group | Afatinib (BIBW2992) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Health Related Quality of Life (HRQOL)
Description: The main analysis of HRQOL questionnaires was to focus on the change in score from baseline in the following scales measured on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 and EORTC QLQ-H&N35:
  * Global Health Status/ Quality of Life (QOL) Scale
  * Pain Scale
  * Swallowing Scale
Time Frame: up to 4 years
Population: as for outcome 1
Arm/Group | Afatinib (BIBW2992) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Safety analysis was based on Treated Set (TS): This analysis set included all patients who received at least one dose of investigational treatment.
Arm/Group | Placebo | Afatinib (BIBW2992)
Serious Adverse Events (participants affected / at risk) | 3/11 | 5/25
Other Adverse Events (participants affected / at risk) | 10/11 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Afatinib (BIBW2992) (N=25)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Afatinib (BIBW2992) (N=25)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 17
Dry mouth (Gastrointestinal disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Localised oedema (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 3
Erythrasma (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Paronychia (Infections and infestations) | 0 | 3
Periodontitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 2
Aspartate aminotransferase decreased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 2
Neutrophil count (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0
Reticulocyte count increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 7
White blood cell count decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 14
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was early terminated by the sponsor along with the global companion trial 1200.131 (NCT01345669), following the recommendation from the external Data Monitoring Committee (DMC) due to futility of 1200.131, but not due to safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.